CLINICAL TRIAL: NCT03918876
Title: Traduzione, Adattamento Transculturale e Misura Delle proprietà Psicometriche Del Questionario "Dance Functional Outcome Survey" (Dfos) in Lingua Italiana
Brief Title: Translation and Psychometric Validation of an Italian Version of the Dance Functional Outcome Survey DFOS-IT
Acronym: DFOS-IT
Status: Completed | Type: Observational
Sponsor: Angela Contri (Other)
Responsible Party: Sponsor-Investigator, Angela Contri, Principal Investigator, University of Bologna
Organization: University of Bologna (Other)
Other Study IDs: 71267
Record Dates: First submitted 2019-04-13; First posted 2019-04-18 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Injuries; Musculoskeletal Pain; Low Back Pain; Lower Limb Injury; Limitation, Mobility; Health Impairment
Keywords: dance; health; ballet; musculoskeletal injury; SF-36; wellness; dance medicine
MeSH Terms: conditions — Wounds and Injuries; Musculoskeletal Pain; Low Back Pain; Leg Injuries; Mobility Limitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healty Dancers: Healthy adult dancers
- Injured Dancers: Injured adult dancers

SUMMARY:
Study Design: Evaluation of the psychometric properties of a translated, culturally adapted questionnaire.

Objective: Translating, culturally adapting, and validating the Italian version of the Dance Functional Outcome Survey (DFOS-IT), allowing its use with Italian-speaking dancers to evaluate their musculoskeletal health and wellbeing inside and outside Italy.

Summary of Background Data: Musculoskeletal injuries are a phenomenon of huge prevalence and has been a major focus within peer-reviewed literature since the 1980s.

Growing attention is devoted to standardized outcome measures to improve interventions for injured dancers.

A translated form of the DFOS, the only existing outcome measure that focus on the unique functional requirements of dancers, has never been validated within the Italian dancers population.

DETAILED DESCRIPTION:
The DFOS is a dance-specific, lower extremity and low back functional outcome measure, the first and only existing at the moment.

The DFOS-IT questionnaire will be developed involving forward-backward translation, a final re-evaluation made by a representative multidisciplinary expert committee and the realization of a prefinal version to establish a proper correspondence with the original English latest version.

A factor analysis and analyses of internal consistency, construct validity, internal responsiveness and sensitivity will be conducted. The reliability will be measured for internal consistency (Cronbach α) and a factor analysis will be applied to analyse the internal structure. The divergent validity will be measured by comparing the data obtained from the compilation of the DFOS-IT with those of the SF-36 to evaluate the psychometric properties and the equivalence of the results adapted to the Italian language and culture.

The validation of the psychometric properties of the instrument will start after it will been administered digitally, via a link to a website built using LimeSurvey, an application based on a MySQL database that allows the realization of online surveys, to a sample population of at least 140 dancers (10 subjects for each item of DFOS-IT) professionals or pre-professionals of age recruited through companies, professional academies, dance high schools and health professionals working with dancers. Through this link, from the time it will be online up to 30 September 2019, the dancers who will give their informed consent to their voluntary participation, will be able to access the online questionnaire.

Upon enrollment, dancers will answer a demographics questionnaire, the DFOS-IT, and the SF-36. If they will take part in the reliability portion, then they filled out the DFOS-IT a second time within 4 to 9 days and, if in the responsiveness testing, a third time after 4-months.

For the statistical analysis standard psychometric techniques will be used, such as reliability assessments, convergent and discriminant validity tests of each item and of the construct in its entirety, empirical validity tests in relation to the clinical status and formal tests to assess their accuracy to ends to test the hypotheses.

The investigators hypothesize to be able to reproduce a tool that reflects the characteristics of the DOFS in the original language and therefore it will prove to have, even in its Italian version, an acceptable psychometric performance as an outcome and screening measure for dancers. The DFOS-IT will show to be a useful tool to monitor both healthy state and functional limitation following lower extremity or low back injury in adult ballet and modern dancers.

ELIGIBILITY:
For all dancers, inclusion criteria :

* A minimum of 3 years of dance training (classical, contemporary, modern-jazz ..)
* An Intermediate to expert skill level
* 18 years of age or older

For healthy dancers subgroup, inclusion criteria:

- No low back or lower extremity injury in the previous 3 months.

For injured dancers subgroup, inclusion criteria:

- at least one low back or lower extremity injury in the previous 3 months.

For all dancers exclusion criteria:

* Non-Italian speaking
* Pregnancy
* Current active disease processes other from a musculoskeletal injury in the low back or lower extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy and injured adult dancers
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2019-05-11 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Dance Functional Outcome Score | 1 day
  Self-reported functional outcome questionnaire for ballet and modern dance populations, applicable to musculoskeletal injuries of the low back and lower extremities. The 14-question DFOS assesses the dancer's ability in areas of activities of daily living (ADL, 40 points) and dance technique (technique, 50 points). Total score from 0 to 90, subscore Activities of daily living 40, Technique 50. Higher scores represent better outcomes. Total points are normalized to a percentage, with 100% representing full function without limitations.
Validate the Italian translation of the DFOS | 1 day
  The score between the DFOS-IT versus the italian validated version of the SF-36 will be compared

SECONDARY OUTCOMES:
DFOS-IT test-retest reliability | Baseline - Between Day 4 and 30
  Assess DFOS-IT test-retest reliabilty in adult dancers with and without musculoskeletal injury to the low back or lower extremities. Test-retest reliability will be assessed with 1 group (including "healthy" and "injured" dancers), 2 measurements (test-retest), with an effect size change of 0.25, power of 0.95, and a significance level of α = .05. Test-retest reliability analysis separately will compare combined, healthy, and injured groups for the DFOS total score and ADL and technique subscores using the intraclass correlation coefficient. The ICC values of 0.49 or less will be considered low, 0.50 to 0.69 moderate, 0.70 to 0.89 high, and 0.90 to 1.00 very high.
DFOS-IT construct validity | Mid December 2019
  Assess DFOS-IT construct validity in with 1 group (adult dancers with and without musculoskeletal injury to the low back or lower extremities), with an effect-size change of 0.25, power of 0.95, and a significance level of α = .05.
DFOS-IT factor analysis and internal consistency | Mid December 2019
  Assess DFOS-IT factor analysis and internal consistency in adult dancers with and without musculoskeletal injury to the low back or lower extremities. Cronbach's alpha will be calculate to estimate internal item consistency.
DFOS-IT sensitivity | Mid December 2019
  Assess DFOS-IT sensitivity in adult dancers with and without musculoskeletal injury to the low back or lower extremities. To conduct sensitivity analyses in the healthy group and injured group, the researchers will conduct a t test for equal variances not assumed and a significant Levene test.
DFOS-IT Internal responsiveness | After 4 months from the first submission
  participants are classified as 'improved' (injured at T0 and healthy at T4mo), 'worsened' (healthy at T0 and injured at T4mo) or 'no change' (health status unchanged from T0 to T4mo). We will examine differences in DFOS-IT and SF-36 scores across 3-time-points using repeated-measures ANOVA. Internal responsiveness was defined using SEM, minimal detectable change at the 95%CI, standardized response mean and effect size and calculated for all DFOS-IT scores, SF-36 PCS and MCS.
DFOS-IT Floor and Ceiling Effects | Mid December 2019
  Assess DFOS-IT Floor and Ceiling Effects in the injured group

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, PT, MSc, Study Chair — University of Bologna; Giorgio Breda, PT, OMT, Study Director — University of Bologna
Locations (1):
- Unità Operativa di Medicina del Lavoro AOU Sant'Orsola-Malpighi, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bronner S, Chodock E, Urbano IER, Smith T. Psychometric Properties of the Dance Functional Outcome Survey (DFOS): Reliability, Validity, and Responsiveness. J Orthop Sports Phys Ther. 2019 Feb;49(2):64-79. doi: 10.2519/jospt.2019.8247. Epub 2018 Jul 27. PMID 30053790
- [Result] Bronner S, Urbano IR. Dance Functional Outcome Survey: Development and Preliminary Analyses. Sports Med Int Open. 2018 Nov 28;2(6):E191-E199. doi: 10.1055/a-0729-3000. eCollection 2018 Nov. PMID 30539138
- [Result] Smith TO, Davies L, de Medici A, Hakim A, Haddad F, Macgregor A. Prevalence and profile of musculoskeletal injuries in ballet dancers: A systematic review and meta-analysis. Phys Ther Sport. 2016 May;19:50-6. doi: 10.1016/j.ptsp.2015.12.007. Epub 2016 Jan 5. PMID 27080110
- [Result] Swain CTV, Bradshaw EJ, Ekegren CL, Whyte DG. The Epidemiology of Low Back Pain and Injury in Dance: A Systematic Review. J Orthop Sports Phys Ther. 2019 Apr;49(4):239-252. doi: 10.2519/jospt.2019.8609. Epub 2019 Jan 18. PMID 30658051
- [Result] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835
- [Result] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Result] Vassallo AJ, Trevor BL, Mota L, Pappas E, Hiller CE. Injury rates and characteristics in recreational, elite student and professional dancers: A systematic review. J Sports Sci. 2019 May;37(10):1113-1122. doi: 10.1080/02640414.2018.1544538. Epub 2018 Nov 27. PMID 30481111
- [Derived] Contri A, Breda G, Vanti C, Pillastrini P, Bronner S. The Dance Functional Outcome Survey: Cultural Adaptation and Psychometric Validation in Italian (DFOS-IT). Med Probl Perform Art. 2021 Sep;36(3):150-162. doi: 10.21091/mppa.2021.3018. PMID 34464961